CLINICAL TRIAL: NCT06806436
Title: Patients' Satisfaction in Thoracic Surgery Inpatients At the Manmohan Cardio-Thoracic Vascular and Transplant Centre: a Cross-sectional Survey
Brief Title: Patients' Satisfaction in Thoracic Surgery Inpatients
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ishwor Thapaliya, Mr., Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 409(6-11)E2
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Thoracic Diseases
MeSH Terms: conditions — Thoracic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Patient satisfaction is considered a subjective indicator of the quality of care provided during a hospital course. Identifying the factors that affect patient satisfaction across remains essential. Recognizing the growing importance of this metric in assessing medical performance, this study aimed to evaluate the satisfaction and associated factors among inpatients of the thoracic surgery unit of a tertiary care government hospital in Nepal.

DETAILED DESCRIPTION:
A cross-sectional analysis of satisfaction levels was conducted among 122 patients consecutively admitted to the Thoracic Surgery unit. Data were collected by interview using a questionnaire of 23 domains scored on a 4-point Likert scale, adapted from the Health Consumer Assessment of Healthcare Providers and Systems (HCAHPS) survey. Descriptive and inferential statistics (independent t-test and Chi-square test) were used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* all patients (or the guardian if the patient was less than 18 years, or could not consent for some reason) admitted to the study site during the study period

Exclusion Criteria:

* refusing to participate, who were hospital staff or their close family members, and those who could not be contacted for interview

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients admitted to the study site during the study period
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Scores of different domains of care received from nurses, doctors and hospital environment | upto 48 hours after discharge
  to assess the satisfaction of inpatients and the factors affecting them in the Thoracic Surgery Service

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan Sapkota, MBBS, MS, Mch, Study Director — Institute of Medicine
Locations (1):
- Institute of Medicine, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) to be shared will include de-identified datasets containing [Patient demographics, clinical characteristics, surgical outcomes, and satisfaction with care apart from patient identifiers]. These datasets will exclude any information that could directly or indirectly identify participants to ensure confidentiality. Summary statistics and study-related documentation, such as the study protocol, statistical analysis plan, and data dictionary, will also be shared.
Supporting Information: Study Protocol, ICF
Time Frame: It will be made available starting after publication of the study results and will remain accessible for 5 years following the initial release date.
Access Criteria: Access to the IPD and supporting information will be granted to researchers upon reasonable request, provided that their proposed use aligns with the study objectives or contributes to furthering knowledge in the field. Researchers must submit a formal request detailing their research goals and sign a data-sharing agreement ensuring data confidentiality and appropriate use. Requests can be made by contacting corresponding or primary author.
  URL to be provided once the data-sharing policy is established.